CLINICAL TRIAL: NCT00089297
Title: Phase II Evaluation of Cetuximab (C225) Combined With Induction Paclitaxel and Carboplatin Followed by C225, Paclitaxel, Carboplatin, and Radiation for Stage III/IV Operable Squamous Cancer of the Head and Neck
Brief Title: Cetuximab, Chemotherapy, and Radiation Therapy for Operable Stage III or IV Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000378194; U10CA021115 (NIH); E2303 (Other: Eastern Cooperative Oncology Group)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Results first posted 2013-03-11 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Cancer
Keywords: Stage III head and neck cancer; Stage IV head and neck cancer; Cetuximab; Paclitaxel; Carboplatin
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cetuximab; Carboplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetuximab/Paclitaxel/Carboplatin (Experimental): Induction: Cetuximab (C225) 400 mg/m2 at wk 1 then 250 mg/m2 for 5 weeks. Paclitaxel (P) 90 mg/m2 IV and carboplatin (C) AUC = 2 IV were given weekly.
  Restaging biopsy of primary site scheduled at wk 7. Concurrent chemoradiation: Radiation therapy at 200cGy/d/5 wks for a total of 50Gy and C225 at 250 mg/m2/wk. P following C225 at 30 mg/m2/wk and C following P at AUC = 1/week. Patients with a negative biopsy continued concurrent therapy to complete radiation (68-72Gy).
  Restaging biopsy of primary site: Patients with positive biopsy at wk 7 or patients without a clinical complete response at the primary site after induction therapy had re-biopsy at wk 14. If the biopsy was negative, the patients continued concurrent therapy to complete radiation (68-72 Gy). If positive, resection of the primary site was done.
  Additional concurrent chemoradiation: C225 at 250mg/m2/wk IV followed by P 30mg/m2/wk IV followed by C AUC = 1/wk and RT for 3 wks.
  Interventions: Biological: Cetuximab; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiation therapy

INTERVENTIONS:
Biological: Cetuximab — Induction: An initial dose of cetuximab (C225) 400 mg/m2 (over 2 hours) was given week 1 only. Then, C225 was administered at dose of 250 mg/m2 (over 1 hour) weekly for 5 weeks.
  Concurrent Chemoradiation (Weeks 9-13): C225 was administered at 250 mg/m2/wk (over 1 hour).
  Restaging Biopsy of Primary Site (Week 14): Patients with positive biopsy of the primary site at week 7 or patients without a clinical complete response at the primary site after induction therapy were scheduled for re-biopsy of the primary site at week 14 after concurrent therapy (50 Gy). If the biopsy were negative after concurrent therapy, the patients were scheduled to continue concurrent therapy to complete radiation (68-72 Gy).
  Additional Concurrent Chemoradiation (weeks 15, 16 and 17): Concurrent therapy was consisted of C225 at 250mg/m2/week IV over 1 hour followed by paclitaxel 30mg/m2/week IV over 1 hour followed by carboplatin AUC = 1/week over 15 minutes and RT for three weeks.
  Other Names: C225; Erbitux
Drug: Carboplatin — Induction Therapy (Week 1-6): The induction chemotherapy starting at week 1 included paclitaxel 90 mg/m2 IV over 1 hour weekly and carboplatin AUC = 2 IV over 30 minutes weekly. The paclitaxel and carboplatin doses were given on the same day, 1 hour after C225 dose was administered. For paclitaxel and carboplatin therapy, rounding of doses (to next decimal if above 0.5 and to lower decimal if below 0.5) was permitted.
  Concurrent Chemoradiation (Weeks 9-13): Concurrent chemotherapy was consisted of paclitaxel following cetuximab at 30 mg/m2/wk (over 1 hour) and carboplatin following paclitaxel at AUC = 1/week (over 15 minutes).
  Additional Concurrent Chemoradiation (weeks 15, 16 and 17): Concurrent therapy was consisted of C225 at 250mg/m2/week IV over 1 hour followed by paclitaxel 30mg/m2/week IV over 1 hour followed by carboplatin AUC = 1/week over 15 minutes and RT for three weeks.
  Other Names: Paraplatin; Paraplatin-AQ
Drug: Paclitaxel — Induction Therapy (Week 1-6): The induction chemotherapy starting at week 1 included paclitaxel 90 mg/m2 IV over 1 hour weekly and carboplatin AUC = 2 IV over 30 minutes weekly. The paclitaxel and carboplatin doses were given on the same day, 1 hour after C225 dose was administered. For paclitaxel and carboplatin therapy, rounding of doses (to next decimal if above 0.5 and to lower decimal if below 0.5) was permitted.
  Concurrent Chemoradiation (Weeks 9-13): Concurrent chemotherapy was consisted of paclitaxel following cetuximab at 30 mg/m2/wk (over 1 hour) and carboplatin following paclitaxel at AUC = 1/week (over 15 minutes).
  Additional Concurrent Chemoradiation (weeks 15, 16 and 17): Concurrent therapy was consisted of C225 at 250mg/m2/week IV over 1 hour followed by paclitaxel 30mg/m2/week IV over 1 hour followed by carboplatin AUC = 1/week over 15 minutes and RT for three weeks.
  Other Names: Taxol
Radiation: Radiation therapy — Concurrent Chemoradiation (Weeks 9-13): Radiation was given at 200cGy/d/5 weeks for a total dose of 50Gy (5000 cGy). Patients with a negative initial biopsy at week 7 were scheduled to continue concurrent therapy to complete radiation (68-72Gy).
  If the biopsy was negative after concurrent therapy, the patients were scheduled to continue concurrent therapy to complete radiation (68-72 Gy).
  Additional Concurrent Chemoradiation (weeks 15, 16 and 17): Concurrent therapy was consisted of C225 at 250mg/m2/week IV over 1 hour followed by paclitaxel 30mg/m2/week IV over 1 hour followed by carboplatin AUC = 1/week over 15 minutes and RT for three weeks.

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving cetuximab with combination chemotherapy and radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving cetuximab after surgery may kill any tumor cells that remain.

PURPOSE: This phase II trial is studying how well giving cetuximab together with combination chemotherapy and radiation therapy works in treating patients who are undergoing surgery for stage III or stage IV head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effect of induction therapy comprising cetuximab, paclitaxel, and carboplatin followed by chemoradiotherapy comprising cetuximab, paclitaxel, carboplatin, and radiotherapy and maintenance therapy comprising cetuximab on 1-year event-free survival (freedom from surgery at the primary site and freedom from recurrence and death) in patients with stage III or IV operable squamous cell cancer of the head and neck.

Secondary

* Determine the pathologic antitumor response at the primary site in patients treated with this regimen.
* Determine disease-free and overall survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine local/regional and distant failure rates in patients treated with this regimen.
* Determine the effect of this treatment regimen on selective biologic pathways, total and phosphorylated epidermal growth factor receptor, ERK/MAPK, and P13K/AKT in these patients.

OUTLINE: This is a multicenter study.

* Induction therapy (weeks 1-6): Patients receive cetuximab IV over 1-2 hours, paclitaxel IV over 1 hour, and carboplatin IV over 30 minutes on days 1, 8, 15, 22, 29, and 36.

During week 7 or 8, patients undergo biopsy and evaluation of the primary site. Patients then proceed to chemoradiotherapy.

* Chemoradiotherapy (weeks 9-13): Patients receive cetuximab IV over 1 hour, paclitaxel IV over 1 hour, and carboplatin IV over 15 minutes on days 57, 64, 71, 78, and 85. Patients also undergo radiotherapy once daily, 5 days a week, on weeks 9-13.

Patients with a positive biopsy at week 7 or 8 or persistent tumor at the primary site after induction therapy undergo a second biopsy after chemoradiotherapy at week 14. Patients with a negative biopsy at week 7 or 8 who achieve a complete clinical and pathological response at the primary site OR patients whose biopsy becomes negative at week 14 receive an additional 3-weeks of chemoradiotherapy beginning at week 15. Patients receive cetuximab, carboplatin, and paclitaxel as in chemoradiotherapy (as outlined above) on days 99, 106, and 113. Patients also undergo radiotherapy once daily, 5 days a week, for 3 weeks (weeks 15-17). Patients with N1-N3 disease undergo neck dissection in weeks 20-21.

Patients with a positive biopsy at week 14 do not receive additional chemoradiotherapy, but rather undergo surgical resection of the primary site in weeks 18-19. Patients with N1-N3 disease also undergo neck dissection at this time.

* Maintenance therapy: Beginning after completion of surgery and/or chemoradiotherapy, patients receive cetuximab IV over 1 hour once weekly for 6 months in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ACTUAL ACCRUAL: A total of 74 patients were accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Locally advanced (Stage III/IV), but potentially operable squamous cancer of the head and neck (exclude nasopharynx). Primary site biopsies must have had proven for cancer, nodal status, confirmed by clinical and pathologic exam with fine needle aspiration cytology recommended.
* ECOG performance status 0 - 1.
* Adequate laboratory index (ANC > 1500/mm3, platelets > 100,000/mm3, creatinine 1.5mg/dl, bilirubin 1.5mg/dl) completed within 4 weeks prior to registration.
* Surgical resectability:

  * Included patients with operative stage III/IV disease, high likelihood of achieving R0 resection (complete resection with clean margins indicating NO residual cancer).
* Measurable disease, biopsy proven at primary site. Patients with clinically palpable cervical nodes were to have evaluation by CT scan and fine needle aspiration (FNA) confirmation of disease. Patients with non-palpable neck nodes had CT determination. In the absence of clinically palpable nodes, radiographic findings were acceptable.
* At least one objective measurable disease parameter in the primary site or neck.
* Baseline measurements or evaluations must have had obtained within 4 weeks prior to registration in the study.
* Age > 18 years.
* Women of childbearing potential and sexually active males were strongly advised to use an accepted and effective method of contraception.
* Original diagnostic materials must have had submitted for baseline EGFR assessment by the designated laboratory.

EXCLUSION CRITERIA:

* Patients with fixed nodal metastases to spine or carotid artery, patients with invasion of root of tongue, pharyngeal muscle, post pharynx, or vertebral fascia or invasion of laryngeal cartilage into strap muscles or tracheal (>1cm) invasion.
* Prior chemotherapy, surgery radiation or immunotherapy for head and neck cancer.
* Prior malignancies except in situ lobular breast carcinoma, in situ cervical carcinoma, basal cell cancers or previously excised and controlled cutaneous squamous cancer (<200 mm thick) were permitted.
* Significant history of cardiac disease i.e., uncontrolled hypertension, unstable angina, congestive heart failure, or uncontrolled arrhythmias.
* Prior anti-epidermal growth factor receptor antibody therapy or therapy with a tyrosine kinase inhibitor including inhibitors targeting EGFR pathway.
* Prior chimerized or murine monoclonal antibody therapy or known allergy to murine proteins or cremophor EL.
* Pregnant or breast-feeding women. All females of childbearing potential must have had a blood test or urine study within 72 hours of study entry and must not have had started therapy until 5 days after registration was over to rule out pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2005-01-06 (Actual); Primary Completion 2010-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold J. Wanebo, MD, Study Chair — Roger Williams Medical Center

REFERENCES:
- [Result] Wanebo HJ, Ghebremichael M, Burtness B, et al.: Phase II evaluation of cetuximab (C225) combined with induction paclitaxel and carboplatin followed by C225, paclitaxel, carboplatin, and radiation for stage III/IV operable squamous cancer of the head and neck (ECOG, E2303). [Abstract] J Clin Oncol 25 (Suppl 18): A-6015, 302s, 2007.
- [Derived] Wanebo HJ, Lee J, Burtness BA, Ridge JA, Ghebremichael M, Spencer SA, Psyrri D, Pectasides E, Rimm D, Rosen FR, Hancock MR, Tolba KA, Forastiere AA. Induction cetuximab, paclitaxel, and carboplatin followed by chemoradiation with cetuximab, paclitaxel, and carboplatin for stage III/IV head and neck squamous cancer: a phase II ECOG-ACRIN trial (E2303). Ann Oncol. 2014 Oct;25(10):2036-2041. doi: 10.1093/annonc/mdu248. Epub 2014 Jul 9. PMID 25009013

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on December 15, 2004, accrued its first patient on January 6, 2005, and was closed to accrual on February 6, 2006 after accruing 74 patients.
Groups:
- Cetuximab/Paclitaxel/Carboplatin: Induction: Cetuximab (C225) 400 mg/m2 at wk 1 then 250 mg/m2 for 5 weeks. Paclitaxel (P) 90 mg/m2 IV and carboplatin (C) AUC = 2 IV were given weekly.
  Restaging biopsy of primary site scheduled at wk 7. Concurrent chemoradiation: Radiation at 200cGy/d/5 wks for a total of 50Gy and C225 at 250 mg/m2/wk. P following C225 at 30 mg/m2/wk and C following P at AUC = 1/week. Patients with a negative biopsy continued concurrent therapy to complete radiation (68-72Gy).
  Restaging biopsy of primary site: Patients with positive biopsy at wk 7 or patients without a clinical complete response at the primary site after induction therapy had re-biopsy at wk 14. If the biopsy was negative, the patients continued concurrent therapy to complete radiation (68-72 Gy). If positive, resection of the primary site was done.
  Additional concurrent chemoradiation: C225 at 250mg/m2/wk IV followed by P 30mg/m2/wk IV followed by C AUC = 1/wk and RT for 3 wks.
Period: Overall Study
Arm/Group | Cetuximab/Paclitaxel/Carboplatin
Started | 74
Treated | 70
Eligible | 63
Completed | 36
Not Completed | 38
Not completed — Adverse Event | 9
Not completed — Death | 1
Not completed — Withdrawal by Subject | 12
Not completed — Disease progression | 2
Not completed — Ineligible | 11
Not completed — Secondary malignancy | 1
Not completed — IRB approval not ready | 1
Not completed — Non-compliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab/Paclitaxel/Carboplatin
Number analyzed (Participants) | 63
Age, Continuous [Median (Full Range); unit: years] | 57 [31 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 49

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival Rate at 1 Year
Description: Event-free survival rate at 1 year was defined as the proportion of patients who did not have disease progression, primary site surgery, or death after being followed for 1 year.
Time Frame: Assessed at 1 year.
Population: Only eligible patients are included in the analysis.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Cetuximab/Paclitaxel/Carboplatin
Number analyzed (Participants) | 63
proportion of patients | 0.79 [0.69 to 0.89]

2. Secondary Outcome: Proportion of Patients With Objective Response by RECIST
Description: Per RECIST criteria, Complete response (CR)= disappearance of all target and nontarget lesions Partial response (PR)= >=30% decrease in the sum of the longest diameters of target lesions from baseline, and persistence of one or more non-target lesion(s) and/or the maintenance of tumor marker level above the normal limits. Objective response = CR + PR.
Time Frame: Assessed at weeks 7, 14, 18, 20, and then every every 3 months if patient is < 2 years from study entry and every 6 months if patient is 2-5 years from study entry
Population: Only eligible patients are included in this analysis.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Cetuximab/Paclitaxel/Carboplatin
Number analyzed (Participants) | 63
proportion of patients | 0.86 [0.75 to 0.93]

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from registration to documented progression or death without progression. Progression is defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s) or unequivocal progression of existing nontarget lesions.
Time Frame: as for outcome 2
Population: Only eligible patients are included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cetuximab/Paclitaxel/Carboplatin
Number analyzed (Participants) | 63
Months | 47.5 [32.6 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from registration to death of any causes.
Time Frame: Weekly during treatment, and then every every 3 months if patient is < 2 years from study entry and every 6 months if patient is 2-5 years from study entry
Population: Only eligible patients are included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cetuximab/Paclitaxel/Carboplatin
Number analyzed (Participants) | 63
Months | 49.4 [47.5 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

ADVERSE EVENTS:
Time Frame: Assessed weekly while on treatment and for 30 days after the end of treatment.
Arm/Group | Cetuximab/Paclitaxel/Carboplatin
Serious Adverse Events (participants affected / at risk) | 64/70
Other Adverse Events (participants affected / at risk) | 70/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab/Paclitaxel/Carboplatin (N=70)
Allergic reaction (Immune system disorders) | 3
Anemia (Blood and lymphatic system disorders) | 1
Leukocytes, decreased (Investigations) | 28
Lymphopenia (Investigations) | 4
Neutrophils, decreased (Investigations) | 31
Fatigue (General disorders) | 6
Weight loss (Investigations) | 7
Burn (Injury, poisoning and procedural complications) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 8
Radiation dermatitis (Injury, poisoning and procedural complications) | 16
Anorexia (Metabolism and nutrition disorders) | 13
Dehydration (Metabolism and nutrition disorders) | 7
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 20
Esophagitis (Gastrointestinal disorders) | 1
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 2
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 35
Muco/stomatitis (symptom) pharynx (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Infection Gr0-2 neut, bladder (Infections and infestations) | 1
Infection Gr0-2 neut, catheter (Infections and infestations) | 2
Infection Gr0-2 neut, colon (Infections and infestations) | 2
Infection Gr0-2 neut, foreign body (Infections and infestations) | 2
Infection Gr0-2 neut, mucosa (Infections and infestations) | 2
Infection Gr0-2 neut, oral cavity (Infections and infestations) | 2
Infection Gr0-2 neut, pharynx (Infections and infestations) | 2
Infection Gr0-2 neut, skin (Infections and infestations) | 1
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 1
Infection w/ unk ANC wound (Infections and infestations) | 1
Blood bilirubin increased (Investigations) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Creatinine, increased (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Neuropathy-motor (Nervous system disorders) | 1
Esophagus, pain (Gastrointestinal disorders) | 1
Oral cavity, pain (Gastrointestinal disorders) | 4
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Obstruction, airway-larynx (Respiratory, thoracic and mediastinal disorders) | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 3
Thrombosis/thrombus/embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab/Paclitaxel/Carboplatin (N=70)
Anemia (Blood and lymphatic system disorders) | 62
Leukocytes, decreased (Investigations) | 61
Lymphopenia (Investigations) | 5
Neutrophils, decreased (Investigations) | 35
Platelets, decreased (Investigations) | 19
Hypotension (Vascular disorders) | 7
Fatigue (General disorders) | 55
Fever w/o neutropenia (General disorders) | 13
Insomnia (Psychiatric disorders) | 7
Weight loss (Investigations) | 42
Activated partial thromboplastin time prolonged (Investigations) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 16
Alopecia (Skin and subcutaneous tissue disorders) | 45
Nail changes (Skin and subcutaneous tissue disorders) | 8
Pruritus/itching (Skin and subcutaneous tissue disorders) | 11
Rash/desquamation (Skin and subcutaneous tissue disorders) | 24
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 64
Radiation dermatitis (Injury, poisoning and procedural complications) | 44
Anorexia (Metabolism and nutrition disorders) | 28
Constipation (Gastrointestinal disorders) | 26
Dehydration (Metabolism and nutrition disorders) | 7
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 16
Dry mouth (Gastrointestinal disorders) | 50
Dysphagia (Gastrointestinal disorders) | 48
Dyspepsia (Gastrointestinal disorders) | 7
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 51
Nausea (Gastrointestinal disorders) | 31
Taste disturbance (Nervous system disorders) | 21
Vomiting (Gastrointestinal disorders) | 19
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 4
Infection Gr0-2 neut, oral cavity (Infections and infestations) | 6
Infection Gr0-2 neut, ungual (Infections and infestations) | 4
Edema limb (General disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
Alanine aminotransferase increased (Investigations) | 36
Aspartate aminotransferase increased (Investigations) | 31
Blood bilirubin increased (Investigations) | 9
Hypocalcemia (Metabolism and nutrition disorders) | 7
Creatinine, increased (Investigations) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 15
Hypokalemia (Metabolism and nutrition disorders) | 9
Hyponatremia (Metabolism and nutrition disorders) | 4
Trismus (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 8
Depression (Psychiatric disorders) | 14
Neuropathy-sensory (Nervous system disorders) | 24
Dry eye syndrome (Eye disorders) | 4
Ocular surface disease (Eye disorders) | 4
Vision-blurred (Eye disorders) | 4
Head/headache (Nervous system disorders) | 11
Joint, pain (Musculoskeletal and connective tissue disorders) | 12
Muscle, pain (Musculoskeletal and connective tissue disorders) | 12
Neck, pain (Musculoskeletal and connective tissue disorders) | 4
Oral cavity, pain (Gastrointestinal disorders) | 10
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 7
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No